CLINICAL TRIAL: NCT06906978
Title: Single Cell Acute Leukemia Analysis
Acronym: SCALA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RCAPHM25_0039; 2025-A00734-45. (Other: ANSM)
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leucemia
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient with acute myeloid leukemia (Other): Adult patient with acute myeloid for whom an additionnal 20 mL of blood will be collected.
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Procedure: blood sampling — Patients will be seen in hospital as part of their routine care, during which a blood test will be prescribed. On this occasion, an additional 20 mlof blood will be collected for research purposes.

SUMMARY:
Numerous chemotherapy and immunotherapy resistance genes have been identified in cancers in general and acute myeloid leukemia in particular. As a preliminary to this study, the investigators hypothesized the co-expression of these genes in the same cell as a major factor in relapse. This hypothesis was supported in vitro by the study of the evolution of these co-expressions after incubation with chemotherapy drugs. The current study aims to verify this hypothesis by studying the expression of these genes in single-cell samples from relapsed acute myeloid leukemia patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient who has received information about the study and has not expressed opposition,
* Patients who are beneficiaries of a social security plan,
* Patient with relapsed or refractory acute myeloid leukemia, whatever the previous treatment, the therapeutic line and the time between the previous treatment and the relapse.

Exclusion Criteria:

* Persons who do not understand the French language if there is no translator available to translate for them.
* Absence of circulating blastosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
percentage of leukemic blasts coexpressing P-glycoprotein (PGP)-Multidrug resistance-related protein (MRP)+ Glutathione S-transferase (GST)+ anti- B-cell Lymphoma 2 (BLC2) | 36 months
  Preliminary in vitro data show that the percentage of blasts coexpressing PGP+MRP+GST+BCL2 is 15% after in vitro chemotherapy. To verify these data in relapsed/refractory patients, the investigators will evaluate the percentage of patients with in vivo leukemic blasts coexpressing PGP+MRP+GST+BCL2 at >15% post-chemotherapy.

SECONDARY OUTCOMES:
percentage of P-glycoprotein (PGP)-Multidrug resistance-related protein (MRP)+ Glutathione S-transferase (GST)+ anti- B-cell Lymphoma 2 (BLC2) coexpression in leukemic blasts | 36 months
  Mean percentages of PGP+MRP+GST+BCL2 co-expression in leukemic blasts from patients with relapsed or refractory acute myeloid leukemia.

CONTACTS AND LOCATIONS:
Overall Officials: Régis Costello, Professor, Principal Investigator — Assitance Public - Hôpitaux de Marseille

IPD SHARING:
Plan to Share IPD: Undecided